CLINICAL TRIAL: NCT04691167
Title: The Role of Repetitive Trans Cranial-magnetic Stimulation in Craving Reduction Among Opioid Use Disorder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Ahmed Saad, assistant lecturer of Neuropsychiatry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: r-TMS
Record Dates: First submitted 2020-10-21; First posted 2020-12-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind sham-controlled randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1, Active intervention group (Active Comparator)
  Interventions: Device: repetitive trans magnetic stimulation
- group 2, sham controlled group (Sham Comparator)
  Interventions: Device: repetitive trans magnetic stimulation

INTERVENTIONS:
Device: repetitive trans magnetic stimulation — Repetitive Trans-cranial Magnetic Stimulation (rTMS) is a relatively safe and non-invasive method to modulate neuronal activity; rTMS uses alternating magnetic fields in a certain frequency to induce an electric current in the underlying brain tissue.
  Other Names: r-TMS

SUMMARY:
Repetitive Trans-cranial Magnetic Stimulation (rTMS) is a relatively safe and non-invasive method to modulate neuronal activity; rTMS uses alternating magnetic fields in a certain frequency to induce an electric current in the underlying brain tissue.

Administering high frequency rTMS to the left dorsolateral prefrontal cortex is possible to increase brain activity in the stimulated area and to change brain activity in associated regions that are part of the same neural circuit which may reduce craving.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-45 years old
2. Gender: males
3. Opioid Use disorder according to the DSM-5 (early abstinence starting 1 week up to 1 month).

Exclusion Criteria:

1. Presence of other serious mental illness (e.g.; psychotic disorders, bipolar affective disorder, depression with psychotic features).
2. Patients with any other serious medical illness.
3. Previous treatment with repetitive Trans- cranial magnetic stimulation.
4. Patients with contraindications to rTMS as cardiac patient with pacemaker.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
craving severity | 6 weeks
  measure severity of drug craving using craving severity scale, the scale is called brief substance craving scale. a higher outcome is a worse result
heroin craving | 6 weeks
  using the heroin craving questionnaire, a higher score indicates a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: amany haroun, BCH, MD, Study Chair — professor at ain shams university, faculty of medicine

IPD SHARING:
Plan to Share IPD: No